CLINICAL TRIAL: NCT03025490
Title: The Use of Capnography and Integrated Pulmonary Index in the Electrophysiology Laboratory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Covidien Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EPCAPNO-HMO-CTIL
Record Dates: First submitted 2016-11-21; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Capnography; Sedation
Keywords: Capnography; Electrophysiology
MeSH Terms: interventions — Capnography

ARMS (2):
- standard of Care (No Intervention): Patient undergoing sedation, treatment team does not have capnography data available.
- Capnography (Experimental): Patient undergoing sedation, treatment team does have capnography data available.
  Interventions: Device: Capnographic monitoring

INTERVENTIONS:
Device: Capnographic monitoring — Capnographic monitoring is used during the sedation.
  Other Names: Capnography; Integrated Pulmonary Index
  Arms: Capnography

SUMMARY:
The study sets out to assess whether in the context of nurse administered procedural sedation in the electrophysiology suite, the routine use of capnography and Integrated Pulmonary Index results in lower incidence of severe adverse respiratory events.

DETAILED DESCRIPTION:
In the electrophysiology lab, the use of procedural sedation, often by nurses is considered routine and safe.Standard monitoring during these procedures includes continuous Oxygen Saturation (SpO2), Heart Rate and rhythm and interval Respiratory rate and blood pressure.

Capnography allows for continuous monitoring of exhaled carbon dioxide, it is an important tool during anesthesia, providing valuable information on the patient's respiratory status and is standard equipment in most operating rooms. Its use in procedural sedation has increased over the past years as the body of evidence supporting this practice has been growing.

It has been previously shown, use of capnography may allow for earlier detection of respiratory adverse events in various types of procedural sedation. The fall of oxygen saturation can occur very late during an adverse respiratory event, especially if supplemental oxygen is given. Today's procedural sedation in the electrophysiology catheterization lab are more complex, patients are of increasingly older age, have more comorbidities, procedures are lengthier and often require deeper sedation (i.e. during complex ablation procedures).

The use of capnography in the electrophysiology lab has not been addressed thoroughly in the literature. A recent multidisciplinary review of anesthesia in the electrophysiology lab states: "In the obstructive sleep apnea or non-obstructive sleep apnea patient, capnography should ideally be employed throughout the sedation period."…"Capnography appears to be underutilized in the electrophysiology lab, given its omission from electrophysiology literature documenting safety of sedation by non-anesthesiologists" We hypothesize that the routine use of capnography during nurse administered procedural sedations in the electrophysiology lab could aid in detection of early signs of adverse respiratory events, thus allowing early intervention and reduction of these events.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older
2. Patient is scheduled to undergo nurse administered procedural sedation in the electrophysiology laboratory.

Exclusion Criteria:

1. Patient is scheduled for anesthesiology based anesthesia.
2. Patient requires ventilator support at baseline (i.e. intubated patient, Bilevel Positive Airway Pressure or continuous positive airway pressure devices are in use)
3. Patient presents to electrophysiology laboratory with capnography monitoring in place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Sentinel Adverse Respiratory Events (AREs) | One month

SECONDARY OUTCOMES:
Mean time to detection of a Sentinel or Moderate ARE | One month
Rate of Moderate Adverse Respiratory Event | One month
Rate of Minor Adverse Respiratory Event | One month
Rate of Minimal Adverse Respiratory Event | One month
Total rate of Adverse Respiratory Event | One month

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem District, Israel

IPD SHARING:
Plan to Share IPD: No